CLINICAL TRIAL: NCT00551083
Title: A Pilot Efficacy Trial of a Computer Decision Support System Compared to Usual Care for Depression Treatment in Primary Care
Brief Title: Efficacy Study of a Computer Decision Support System to Treat Depression
Acronym: CDSS-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Pfizer (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1143107; R01 MH-164062-01A1
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2007-10-30 (Estimated); Status verified 2007-10

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CDSS-D (Experimental): Computer Decision Support System for Depression (CDSS-D) - This arm provided physicians with a computerized treatment algorithm and a decision support system to treat their patients suffering Major Depressive Disorder
  Interventions: Other: Computerized Decision Support System for Depression (CDSS-D)
- UC (Active Comparator): Usual Care (UC) - This group of physicians treated their patients suffering from Major Depressive Disorder with their standard treatment as usual, and received no algorithm support with regard to treatment decisions
  Interventions: Other: Usual Care (UC)

INTERVENTIONS:
Other: Computerized Decision Support System for Depression (CDSS-D) — The CDSS for depression was based on an up-to-date model of the Texas Medication Algorithm Project that employs the principles of Measurement Based Care (MBC), while at the same time having a user interface for providers that is easy-to-use. MBC is the systematic use of measuring clinical outcomes at routine visits to guide treatment management. These outcomes may include symptoms, side effects, and medication adherence. Recent efforts from the large, multi-site effectiveness study, Sequenced Treatment Alternatives to Relieve Depression (STAR*D), show that a treatment plan guided by MBC is integral in implementing algorithm based care.
  Arms: CDSS-D
Other: Usual Care (UC) — Usual Care was up to the discretion of the study physician and the patient treated. These physicians were provided with up-to-date treatment protocols for depression, but were not instructed to strictly adhere to a treatment algorithm. Therefore, they treated depressed patients as they "usually" would.
  Arms: UC

SUMMARY:
The purpose of this study was designed to test the feasibility and effectiveness of implementing a Computerized Decision Support System for depression (CDSS-D) during acute care in a primary care setting.

DETAILED DESCRIPTION:
The research project was designed to test the feasibility and effectiveness of implementing a Computerized Decision Support System for depression (CDSS-D) during acute care in a primary care setting. The basic experimental design was a two-group, two-site study design. Three different clinics with a total of 4 primary care physicians agreed and provided informed consent and participated in the study. Half of the physicians used the CDSS-D to treat patients with MDD and the other half provided Usual Care (UC) treatment.

The intervention, CDSS-D, incorporated a pre-existing depression treatment algorithm (Texas Medication Algorithm Project for Depression, Trivedi et al) with computer decision support programming, providing the treatment group physicians with a computerized algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged 18 and over
* Met Criteria for Non-Psychotic Major Depressive Disorder
* Had a baseline HRSD-17 score of at least 14

Exclusion Criteria:

* Patients with a current Axis I diagnosis of somatization disorder, anorexia nervosa, bulimia, or obsessive-compulsive disorder
* Patients with current alcohol or substance dependence
* Women with a positive pregnancy test or who are lactating
* Women of child-bearing potential who are not practicing a clinically accepted method of contraception
* Patients with general medical conditions that contraindicate antidepressant medications
* Patient whose clinical status requires inpatient or day hospital treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-03; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in the 17-item Hamilton Rating Scale for Depression (HRSD) Score | 24 weeks

SECONDARY OUTCOMES:
Mean change from baseline on the 16-item Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR-16) | 24 weeks
Mean change from baseline on the 30-item Inventory of Depressive Symptomatology - Clinician's version (IDS-C-30) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar H. Trivedi, M.D., Principal Investigator — University of Texas Southwestern Medical Center

REFERENCES:
- [Derived] Kurian BT, Trivedi MH, Grannemann BD, Claassen CA, Daly EJ, Sunderajan P. A computerized decision support system for depression in primary care. Prim Care Companion J Clin Psychiatry. 2009;11(4):140-6. doi: 10.4088/PCC.08m00687. PMID 19750065